CLINICAL TRIAL: NCT05621811
Title: Double-blind, Randomised, Placebo-controlled, Dose-finding Phase IIb Trial to Evaluate the Efficacy, Safety, and Tolerability of a 12-week-treatment with Naronapride in Adult Participants with At Least Moderate Idiopathic or Diabetic Gastroparesis
Brief Title: Different Doses of Naronapride Vs. Placebo in Gastroparesis
Acronym: MOVE-IT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAT-19/GPX
Record Dates: First submitted 2022-11-03; First posted 2022-11-18 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-08

CONDITIONS: Gastroparesis
Keywords: stomach; diabetes mellitus
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus | interventions — ATI 7505

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Naronapride 10 mg (Experimental)
  Interventions: Drug: Naronapride
- Naronapride 20 mg (Experimental)
  Interventions: Drug: Naronapride
- Naronapride 40 mg (Experimental)
  Interventions: Drug: Naronapride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naronapride — Naronapride is a 5HT-4 agonist
  Arms: Naronapride 10 mg; Naronapride 20 mg; Naronapride 40 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, multicenter, placebo-controlled, comparative phase II dose-finding trial. The trial will be conducted with four treatment groups in the form of a parallel group comparison and will serve to compare oral treatment with daily doses of 10, 20, or 40 mg Naronapride vs. placebo for the treatment of patients with Gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between ≥18 and ≤75 years of age,
* Body Mass Index (BMI) ≥16 and <35 kg/m2 ,
* History of idiopathic or diabetic gastroparesis cardinal symptoms (e.g., nausea, vomiting, early satiety, postprandial fullness, bloating or upper abdominal pain) for ≥3 months,
* Evidence of delayed gastric emptying by 13C-spirulina gastric emptying breath test (GEBT) for solids with gastric emptying T1/2 ≥ 85.33 minutes (≥ 90th percentile of normative data) during the screening phase,
* Average weekly total symptom score of the ANMS GCSI-DD ≥2.0 based on the daily symptom scores recorded for at least 5 of 7 consecutive days in the week prior to Baseline,
* Participants with a type I or type II diabetes mellitus diagnosis must have a controlled diabetes mellitus defined as HbA1c ≤11% under stable antidiabetic medication,
* Exclusion of any mechanical and/or anatomical obstructions, stenosis, structural diseases, or gastric ulcers by upper gastrointestinal endoscopy during screening phase (previous endoscopic results within 12 months are acceptable, if no relevant changes in patient's disease status occurred since that time),
* No evidence of intestinal stenosis as determined by an imaging technique (i.e., either abdominal sonography, Magnetic resonance imaging [MRI] or imaging by computed tomography [CT] during screening phase (previous MRI/CT imaging or sonography results within 12 months are acceptable, if no relevant changes occurred in patient's disease status since that time),

Exclusion Criteria:

* History of major gastrointestinal surgery such as gastric bypass, anti-reflux surgery, gastric per oral endoscopic myotomy (G-POEM), gastrointestinal malignancy, colectomy,
* Intrapyloric botulinum toxin injection within 12 months,
* Gastric stimulator implant,
* Known secondary causes of gastroparesis including but not limited to Parkinson's Disease, cancer, or connective tissue diseases,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index - Daily Diary total score from baseline to week 12 | 12 weeks

CONTACTS AND LOCATIONS:
Locations (20):
- United States (19):
  - Dr Falk Investigational Site, Chula Vista, California
  - Dr Falk Investigational Site, Lomita, California
  - Dr Falk Investigational Site, Clearwater, Florida
  - Dr Falk Investigational Site, Doral, Florida
  - Dr Falk Investigational Site, Hollywood, Florida
  - Dr Falk Investigational Site, Maitland, Florida
  - Dr Falk Investigational Site, Miami, Florida
  - Dr Falk Investigational Site, Viera, Florida
  - Dr Falk Investigational Site, Topeka, Kansas
  - Dr Falk Investigational Site, Crestview Hills, Kentucky
  - Dr Falk Investigational Site, Houma, Louisiana
  - Dr Falk Investigational Site, Marrero, Louisiana
  - Dr Falk Investigational Site, Flint, Michigan
  - Dr Falk Investigational Site, New York, New York
  - Dr Falk Investigational Site, Tulsa, Oklahoma
  - Dr Falk Investigational Site, Philadelphia, Pennsylvania
  - Dr Falk Investigational Site, Cordova, Tennessee
  - Dr Falk Investigational Site, Nashville, Tennessee
  - Dr Falk Investigational Site, Harlingen, Texas
- University of Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No